CLINICAL TRIAL: NCT06911632
Title: MOMENTOUS Study (iMpact Of an Ecg ai ModEl oN The Diagnosis Of pUlmonary hypertenSion)
Brief Title: Multi-site Study of the Clinical Impact of an AI-assisted Approach to Referring Patients With Interstitial Lung Disease for Diagnostic Evaluation of Pulmonary Hypertension
Acronym: MOMENTOUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tempus AI (Industry)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TP-CA-008
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease (ILD)
Keywords: Pulmonary Hypertension; Interstitial lung disease (ILD)
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: An ECG-based AI device, will provide a prediction of a participant's risk of having undiagnosed pulmonary hypertension. Participants with a high risk prediction in the Device group will undergo a transthoracic echocardiogram and a right heart catheterization (RHC). All other participants will receive standard of care treatment.
Masking Description: For participants in the Device group, the risk prediction will be returned to the treating provider whereas the providers will be blinded to the risk predictions for participants in the Control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- High Risk Device (Experimental): The device result will be returned to the treating provider and participants will undergo a study sponsored diagnostic work-up consisting of a transthoracic echocardiogram and an RHC.
  Interventions: Device: ECG-based AI Device - Results Returned to Investigator; Procedure: Echocardiogram and Right Heart Catheterization
- Not High Risk Device (Experimental): The device result will be returned to the treating provider. Participants will continue to be evaluated for PH according to the current standard of care with any diagnostic procedures ordered at the discretion of the treating provider.
  Interventions: Device: ECG-based AI Device - Results Returned to Investigator
- High Risk Control Arm (Other): The device result will not be returned to the treating provider. Participants will continue to be evaluated for PH according to the current standard of care with any diagnostic procedures ordered at the discretion of the treating provider.
  Interventions: Device: ECG-based AI Device - Results Not Returned to Investigator
- Not High Risk Control Arm (Other): The device result will not be returned to the treating provider. Participants will continue to be evaluated for PH according to the current standard of care with any diagnostic procedures ordered at the discretion of the treating provider.
  Interventions: Device: ECG-based AI Device - Results Not Returned to Investigator

INTERVENTIONS:
Device: ECG-based AI Device - Results Returned to Investigator — An ECG-based AI device that predicts undiagnosed PH using data from a 12-lead ECG. Device results will be returned to the Investigators.
  Arms: High Risk Device; Not High Risk Device
Procedure: Echocardiogram and Right Heart Catheterization — Echocardiogram- an ultrasound study of the heart and Right Heart Catheterization- a procedure to measure pressures in the heart
  Arms: High Risk Device
Device: ECG-based AI Device - Results Not Returned to Investigator — An ECG-based AI device that predicts undiagnosed PH using data from a 12-lead ECG. Device results will not be returned to the Investigators.
  Arms: High Risk Control Arm; Not High Risk Control Arm

SUMMARY:
MOMENTOUS is a multi-center, randomized study to prospectively evaluate the performance of an ECG-based AI device to predict whether participants with interstitial lung disease (ILD) are at high risk of undiagnosed pulmonary hypertension.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the use of an ECG-based AI device that may help predict if participants with interstitial lung disease (ILD) are at high risk of undiagnosed pulmonary hypertension (PH). The study seeks to determine whether use of the device increases the rate of new PH diagnoses over a period of 6 months as compared to current standard of care.

The study will recruit participants with ILD from lung disease clinics who will each receive a 12-lead ECG (a test that measures the electrical activity of the heart) following consent. The device will analyze the 12-lead ECG results to identify participants that are at high risk of having undiagnosed PH.

Participants will be randomly assigned to either the Device or Control group. For participants in the Device group investigators will receive the results of the device. In the Control group investigators will not receive the results of the device. Additionally, participants in the Device group identified as "high risk" by the device will receive a transthoracic echocardiogram and a right heart catheterization (RHC). Participants in the Device group who are not high risk and all participants in the Control group will not receive these additional tests as part of the study, but will receive standard of care treatment as determined by their physicians, which may include an echocardiogram or RHC if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of consent
* A known diagnosis of interstitial lung disease
* Willing and able to provide informed consent and undergo all study-specific procedures, including echo and RHC, if required

Exclusion Criteria:

* A known diagnosis of pulmonary hypertension (including patients prescribed a therapy specifically for pulmonary arterial hypertension (PAH))
* A RHC was completed within the previous 1 year or ordered and not yet completed at the time of consent
* LV ejection fraction ≤ 40% on most recent echo or cardiac MRI, if available
* Unclassifiable Tempus PH ECG risk result after up to 2 ECG acquisitions
* A contraindication to RHC exists (for example, mechanical right heart valve)
* Physician decision that if a patient is directed to RHC by the study protocol, the potential risks of RHC outweigh the potential benefits
* There is a severe concomitant illness limiting life expectancy to less than 6 months (at the discretion of the investigator)
* There is a medical or social factor that makes the patient a poor candidate for the study and/or unlikely to be able to comply with the study protocol or complete study procedures (at the discretion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants receiving a new diagnosis of PH within the High risk Device group compared to the High risk Control group. | Through study completion, approximately 6 months
  Mean pulmonary artery pressure (mPAP) > 20 mm Hg and pulmonary vascular resistance (PVR) > 2 Wood units

SECONDARY OUTCOMES:
Proportion of participants receiving a new diagnosis of PH within the Device group compared to the Control group. | Through study completion, approximately 6 months
  mPAP > 20 mm Hg and PVR > 2 Wood units
Proportion of participants receiving a new diagnosis of PH within the High risk Device group compared to the Not high risk Device group. | Through study completion, approximately 6 months
  mPAP > 20 mm Hg and PVR > 2 Wood units

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - Dignity Health - St. Joseph's Hospital and Medical Center-Norton Thoracic Institute, Phoenix, Arizona
  - National Jewish Health, Denver, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois Health, Chicago, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Community Health Network, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Shreveport, Shreveport, Louisiana
  - University of Michigan - Michigan Medicine, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - CHI Health Creighton University Medical Center - Bergan Mercy, Omaha, Nebraska
  - University of Buffalo, Buffalo, New York
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Temple University of The Commonwealth System of Higher Education, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - West Virginia University Hospital, Morgantown, West Virginia